CLINICAL TRIAL: NCT02454296
Title: Paracervical Block for Pain Associated With Laminaria Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Reni Soon, Assistant Professor, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22702
Record Dates: First submitted 2015-05-18; First posted 2015-05-27 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Pain
Keywords: Laminaria
MeSH Terms: conditions — Pain | interventions — Anesthesia, Obstetrical; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paracervical Block with lidocaine (Active Comparator): A paracervical block will be done prior to the placement of laminaria with 1% lidocaine and sodium bicarbonate.
  Interventions: Drug: Paracervical Block with lidocaine
- Sham paracervical block (Sham Comparator): A sham block will be done prior to the placement of laminaria using a capped needle
  Interventions: Drug: Sham paracervical block

INTERVENTIONS:
Drug: Paracervical Block with lidocaine — Performance of paracervical block, using 18 mL of 1% lidocaine buffered with 2 mL 8.4% sodium bicarbonate, prior to laminaria insertion
  Other Names: Paracervical block
  Arms: Paracervical Block with lidocaine
Drug: Sham paracervical block — A capped needle will be placed on the cervix prior to laminaria insertion for purposes of blinding both the participant and research staff assessing outcomes
  Other Names: Sham block; placebo
  Arms: Sham paracervical block

SUMMARY:
To assess if paracervical block is effective at reducing discomfort during placement of intracervical laminaria for pre-operative cervical preparation.

DETAILED DESCRIPTION:
Pre-operative dilation of the cervix with use of osmotic dilators (e.g. laminaria, dilapan-S) is commonly done prior to pregnancy termination to make the procedure safer. This study seeks to assess whether paracervical blocks are effective at reducing pain associated with placement of laminaria. Secondarily, this study will evaluate if paracervical blocks are effective at reducing overall procedural pain and increasing overall patient satisfaction for the intracervical laminaria placement procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-49 years
* Desiring surgical termination of pregnancy or surgical management of a fetal demise
* Treatment plan involves cervical preparation with laminaria
* Participant able to provide informed consent in English and willing to participate in the study

Exclusion Criteria:

* Unable to read/speak/understand English
* Contraindications to receiving lidocaine

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — University of Hawaii
Locations (1):
- University Women's Health Specialists, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grimes DA, Schulz KF, Cates WJ Jr. Prevention of uterine perforation during curettage abortion. JAMA. 1984 Apr 27;251(16):2108-11. PMID 6708260
- [Background] Renner RM, Nichols MD, Jensen JT, Li H, Edelman AB. Paracervical block for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):1030-7. doi: 10.1097/AOG.0b013e318250b13e. PMID 22525915
- [Background] Kan AS, Ng EH, Ho PC. The role and comparison of two techniques of paracervical block for pain relief during suction evacuation for first-trimester pregnancy termination. Contraception. 2004 Aug;70(2):159-63. doi: 10.1016/j.contraception.2004.03.013. PMID 15288222
- [Background] Mercier RJ, Liberty A. Intrauterine lidocaine for pain control during laminaria insertion: a randomized controlled trial. Contraception. 2014 Dec;90(6):594-600. doi: 10.1016/j.contraception.2014.07.008. Epub 2014 Jul 23. PMID 25139724
- [Background] Borgatta L, Roncari D, Sonalkar S, Mark A, Hou MY, Finneseth M, Vragovic O. Mifepristone vs. osmotic dilator insertion for cervical preparation prior to surgical abortion at 14-16 weeks: a randomized trial. Contraception. 2012 Nov;86(5):567-71. doi: 10.1016/j.contraception.2012.05.002. Epub 2012 Jun 6. PMID 22682721
- [Background] Drey EA, Benson LS, Sokoloff A, Steinauer JE, Roy G, Jackson RA. Buccal misoprostol plus laminaria for cervical preparation before dilation and evacuation at 21-23 weeks of gestation: a randomized controlled trial. Contraception. 2014 Apr;89(4):307-13. doi: 10.1016/j.contraception.2013.10.013. Epub 2013 Nov 4. PMID 24560477
- [Background] Goldberg AB, Drey EA, Whitaker AK, Kang MS, Meckstroth KR, Darney PD. Misoprostol compared with laminaria before early second-trimester surgical abortion: a randomized trial. Obstet Gynecol. 2005 Aug;106(2):234-41. doi: 10.1097/01.AOG.0000168629.17326.00. PMID 16055570
- [Background] Prairie BA, Lauria MR, Kapp N, Mackenzie T, Baker ER, George KE. Mifepristone versus laminaria: a randomized controlled trial of cervical ripening in midtrimester termination. Contraception. 2007 Nov;76(5):383-8. doi: 10.1016/j.contraception.2007.07.008. Epub 2007 Oct 4. PMID 17963864
- [Background] Hakim-Elahi E, Tovell HM, Burnhill MS. Complications of first-trimester abortion: a report of 170,000 cases. Obstet Gynecol. 1990 Jul;76(1):129-35. PMID 2359559
- [Background] Blanco LJ, Reid PR, King TM. Plasma lidocaine levels following paracervical infiltration for aspiration abortion. Obstet Gynecol. 1982 Oct;60(4):506-8. PMID 7121936
- [Derived] Soon R, Tschann M, Salcedo J, Stevens K, Ahn HJ, Kaneshiro B. Paracervical Block for Laminaria Insertion Before Second-Trimester Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2017 Aug;130(2):387-392. doi: 10.1097/AOG.0000000000002149. PMID 28697113
- See also: Summary of lidocaine drug information — http://www.pdr.net/drug-summary/xylocaine-xylocaine-with-epinephrine-xylocaine-mpf-xylocaine-mfp-with-epinephrine?druglabelid=2543&id=2148

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from May 2015 to Dec 2015 at two of the faculty practice offices of the University of Hawaii Department of OB/gyn.
Period: Overall Study
Arm/Group | Paracervical Block With Lidocaine | Sham Paracervical Block
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paracervical Block Group: Participants in this arm received a paracervical block consisting of 18 ml 1% lidocaine and 2 ml 8.4% sodium bicarbonate prior to the placement of laminaria.
- Sham Block Group: Participants in this arm had a 20 ml syringe with a capped needle applied to the cervix.
- Total: Total of all reporting groups
Arm/Group | Paracervical Block Group | Sham Block Group | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.80 (6.12) | 29.81 (6.92) | 27.85 (6.77)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Females | 20 | 21 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were allowed to mark more than one race
  Participants
    White/Caucasian | 5 | 7 | 12
    Black/African American | 1 | 0 | 1
    Asian | 5 | 9 | 14
    Native Hawaiian/Pacific Islander | 10 | 10 | 20
    Hispanic/Latina | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Pain After Placement of Laminaria (100 mm Visual Analog Scale)
Description: We asked the participant to rate her pain on a 100 mm Visual Analog Scale (VAS) immediately after laminaria was placed. The VAS is a validated measure of pain where 0=no pain and 100=worst pain ever felt.
Time Frame: Measured within 10 seconds after placement of laminaria
Measure: Median (Inter-Quartile Range); unit: units on a scale (100 mm VAS)
Arm/Group | Paracervical Block With Lidocaine | Sham Paracervical Block
Number analyzed (Participants) | 20 | 21
units on a scale (100 mm VAS) | 13 [2 to 39] | 54 [27 to 61]
Statistical Analysis 1: Comparison: Paracervical Block With Lidocaine vs Sham Paracervical Block; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Satisfaction With Overall Pain Control (100 mm Visual Analog Scale)
Description: Patients rated their satisfaction with overall pain control on the 100 mm VAS, with 0 as not satisfied at all and 100 as completely satisfied
Time Frame: 15 minutes post-operatively
Measure: Median (Inter-Quartile Range); unit: units on a scale (100 mm VAS)
Arm/Group | Paracervical Block Group | Sham Block Group
Number analyzed (Participants) | 20 | 21
units on a scale (100 mm VAS) | 95 [78 to 100] | 70 [44 to 90]
Statistical Analysis 1: Comparison: Paracervical Block Group vs Sham Block Group; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Paracervical or Sham Block Pain
Description: Participants reported her pain level on the 100 mm Visual Analog Scale (VAS) within 10 seconds after she received either the paracervical block or the sham block. The VAS is a validated measure of pain where 0=no pain and 100=worst pain ever felt.
Time Frame: Within 10 seconds after receiving paracervical or sham block
Measure: Median (Inter-Quartile Range); unit: units on a scale (100 mm VAS)
Arm/Group | Paracervical Block Group | Sham Block Group
Number analyzed (Participants) | 20 | 21
units on a scale (100 mm VAS) | 14 [6 to 31] | 27 [6 to 41]
Statistical Analysis 1: Comparison: Paracervical Block Group vs Sham Block Group; Test type: Superiority or Other; p = 0.34, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Paracervical Block With Lidocaine | Sham Paracervical Block
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

LIMITATIONS AND CAVEATS:
1. Overall pain scores lower than in other published studies - speaks to generalizability
2. Paracervical block formulation might not be what is commonly used elsewhere
3. 76% of participants were able to correctly guess their group allocation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No